CLINICAL TRIAL: NCT06323395
Title: Multi-centre, Randomised,Parallel-group, Controlled (Placebo), Double-blind Study to Evaluate the Efficacy, Ocular Tolerability and Safety of Vizol S Lipid Balance in the Adult Patient Population With Moderate to Severe Dry Eye for up to 30 Days
Brief Title: Vizol S Lipid Balance Efficacy and Safety Study in Patients With Dry Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jadran Galenski laboratorij d.d. (Industry)
Collaborators: Poseidon CRO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: JGL-DED-VIZ-SLB 21
Record Dates: First submitted 2024-03-07; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-12

CONDITIONS: Dry Eye Disease
Keywords: keratoconjunctivitis sicca (KCS); KCS; DED; dry eye syndrome; moderate dry eye disease; severe dry eye disease; evaporative DED
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca

STUDY DESIGN:
Intervention Model Description: Multi-centre, randomised, parallel-group, controlled (placebo), double-blind study
Who Masked: Participant, Care Provider, Investigator
Masking Description: As the clinical trial will be conducted in a double-blind way, both investigators and patients will be blind with respect to the treatment administered. For the purpose of individual unblinding of a patient's treatment the investigator will receive a sealed emergency envelope for each patient containing the treatment code (Only in case of medical emergency it is permitted to open the emergency envelope).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vizol S LIPID BALANCE (Experimental): topical administration of 1 drop of Vizol S LIPID BALANCE in each eye 4 times a day for 30 days
  Interventions: Drug: Vizol S LIPID BALANCE eye drops
- ophthalmic saline eyedrops (Placebo Comparator): topical administration of 1 drop of ophthalmic saline eye drops matching Vizol S LIPID BALANCE in each eye 4 times a day for 30 days
  Interventions: Drug: ophthalmic saline eye drops

INTERVENTIONS:
Drug: Vizol S LIPID BALANCE eye drops — 1 drop 4 times a day
  Other Names: Test
  Arms: Vizol S LIPID BALANCE
Drug: ophthalmic saline eye drops — 1 drop 4 times a day
  Other Names: Placebo
  Arms: ophthalmic saline eyedrops

SUMMARY:
The clinical investigation was intended to investigate the efficacy, ocular tolerability and safety of Vizol S Lipid Balance, a new eye drops, emulsion developed by JADRAN - GALENSKI LABORATORIJ d.d., in patients with moderate to severe evaporative DED after a treatment for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* use of eyelid hygiene for at least 14 days prior to screening
* diagnosis of moderate to severe dry eye disease (DED), with an Ocular Surface Disease Index (OSDI) score ≥23
* Tear Film Break-Up Time (TFBUT) <10 seconds in one or both eyes
* Meibomian gland expression of grade 2 or higher in both eyes
* written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the patients participating in the clinical trial

Exclusion Criteria:

* intolerance or hypersensitivity to any component of the Investigational Product (IPs)
* ocular or intraocular surgery or serious ocular trauma ≤6 months before enrolment
* current punctal occlusion of any type
* use of concomitant topical ocular medications within 24 hours prior to first intended administration of the IPs (except for artificial tears or lubricants; previously used artificial tears or lubricants must be suspended for the duration of the study)
* use of systemic medications that may contribute to dry eye (unless on a stable regimen for ≥30 days before screening and throughout the study)
* current or previous topical treatment of the eye with antibiotics, steroids or cyclosporin A within the last four weeks
* ocular or systemic infections or conditions (e.g., epithelial herpes simplex keratitis, vaccinia, varicella, or mycobacterial infection, fungal disease, iritis) or other relevant ocular pathology judged by the investigator that preclude safe administration of the IPs
* use of contact lenses within 1 week before screening and throughout the study
* active ocular disease other than DED or any other acute or chronic disease which may interfere with the aims of the clinical trial
* history of severe allergies or multiple drug allergies unless it is judged as not relevant for the clinical trial by the investigator
* diagnosis of Corona Virus Disease (COVID-19) within the last 14 days prior to individual enrolment of the patient
* contact to persons in international risk areas for COVID-19 as defined by the Institute of Public Health of Serbia within the last 14 days prior to individual enrolment of the patient
* known direct contact with insufficient protection to persons with diagnosis of COVID-19 within the last 14 days prior to individual enrolment upon reporting of the patient
* history of or current drug or alcohol dependence
* participation in an investigational drug or device study ≤30 days before screening
* positive pregnancy test at screening examination
* pregnant or lactating women
* female patients who do not agree to apply highly effective contraceptive methods (highly effective contraceptive methods are defined in chapter 13.2.1)
* patients suspected or known not to follow instructions
* patients who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Mean change in the tear film break-up time (TFBUT) from Visit 1 (baseline) to Visit 3 (day 30) | baseline, week 2 follow-up and week 4 follow-up
  Tear film break-up time (TFBUT) will be assessed at each visit following the instillation of fluorescein solution into the eye. Fluorescein will be instilled at the outer canthus to avoid ocular surface damage, with the excess saline on the strip shaken off, or a reduced area fluorescein strip used. Viewing will take place between 1 and 3 min after instillation.
  Three measurements per eye will be performed and the mean value documented and used for evaluation.

SECONDARY OUTCOMES:
Mean change in the tear film break-up time (TFBUT) from Visit 1 (baseline) to Visit 2 (day 15) | baseline and week 2 follow-up
  Tear film break-up time (TFBUT) will be assessed following the instillation of fluorescein solution into the eye. Fluorescein will be instilled at the outer canthus to avoid ocular surface damage, with the excess saline on the strip shaken off, or a reduced area fluorescein strip used. Viewing will take place between 1 and 3 min after instillation.
  Two measurements per eye will be performed and the mean value documented and used for evaluation
percent (%) change in the tear film break-up time (TFBUT) from Visit 1 (baseline) to Visit 2 (day 15) and from Visit 1 (baseline) to Visit 3 (day 30) | baseline and week 2 follow-up; baseline and week 4 follow-up
  Tear film break-up time (TFBUT) will be assessed following the instillation of fluorescein solution into the eye. Fluorescein will be instilled at the outer canthus to avoid ocular surface damage, with the excess saline on the strip shaken off, or a reduced area fluorescein strip used. Viewing will take place between 1 and 3 min after instillation.
  Two measurements per eye will be performed and the mean value documented and used for evaluation
Mean change in ocular surface staining score (total corneal and total conjunctival staining score) from Visit 1 (baseline) to Visit 3 (day 30) | baseline, week 2 follow-up and week 4 follow-up
  Ocular surface staining of five corneal regions and six conjunctival regions will be observed at each visit by slit-lamp examination after instillation of fluorescein respectively.
  Surface staining will be scored as 0 (normal, no staining), 1 (mild, superficial stippling or macropunctate staining), 2 (moderate, macropunctate staining with some coalescent areas), or 3 (severe, numerous coalescent macropunctate areas or patches). Scores will be summed to yield total corneal and total conjunctival staining scores for each eye.
Mean change in OSDI score from Visit 1 (baseline) to Visit 3 (day 30) | baseline, week 2 follow-up and week 4 follow-up
  Symptoms of DED will be assessed using the Ocular Surface Disease Index (OSDI) questionnaire at each visit.
  The 12-item OSDI questionnaire scores range from 0 to 100, it contains 3 ocular symptom questions, 6 vision-related function questions, and 3 environmental trigger questions. Each question score ranges from 0 ("none of the time") to 4 ("all of the time"). The total score is calculated based on the following formula:
  Total score: OSDI = ([sum of scores for all questions answered*100]/[total number of questions answered*4])
Mean change in Meibomian gland expression from Visit 1 (baseline) to Visit 3 (day 30) | baseline, week 2 follow-up and week 4 follow-up
  Meibomian gland expression will be observed by slit-lamp examination. Glands will be expressed from the temporal to the nasal aspect using a cotton-tipped applicator. Five glands in each area of the lower lid (nasal, central, temporal) will be examined.
  Expressed meibum (across all glands) will be classified as follows: clear, easily expressed (grade 0), cloudy, mild pressure (grade 1), cloudy, > moderate pressure (grade 2), meibum not expressed, with hard pressure (grade 3).

OTHER OUTCOMES:
The presence of Adverse Event/ /Serious Adverse Event (AE/ /SAE) throughout the investigation period | baseline, week 2 follow-up and week 4 follow-up
  The patients will be asked to report any Pre-Treatment Sign and Symptom/Adverse Events (PTSS/AEs) spontaneously.
BCVA | baseline, week 2 follow-up and week 4 follow-up
  Best corrected visual acuity (BCVA) will be assessed at each visit. BCVA assessment will be at 4 meters using an ETDRS chart (The Early Treatment Diabetic Retinopathy Study Group). Results will be calculated as logMAR scores.
Frequency of ocular signs | baseline, week 2 follow-up and week 4 follow-up
  Ocular signs will be assessed by slit-lamp examination at all study visits. The following signs will be assessed:
  * active inflammation or significant structural change or discharge (eyelids and conjunctiva);
  * active inflammation or active structural change, including focal scarring and fine deposition (cornea);
  * active inflammation (iris and anterior chamber);
  * level of lens opacity, pseudophakia, or aphakia (lens, with an emphasis on the visual axis)

CONTACTS AND LOCATIONS:
Overall Officials: D. Veselinović, prof. dr., Principal Investigator — Specialized clinic for eye desease - klinika Veselinović
Locations (2):
- Serbia (2):
  - Special eye hospital - Beogradski oftalmološki centar, Belgrade
  - Specialized clinic for eye desease - klinika Veselinović, Niš

IPD SHARING:
Plan to Share IPD: No
Individual Participant Datas (IPDs) are available to the Health Authorities on a request

REFERENCES:
- [Result] Wolffsohn JS, Arita R, Chalmers R, Djalilian A, Dogru M, Dumbleton K, Gupta PK, Karpecki P, Lazreg S, Pult H, Sullivan BD, Tomlinson A, Tong L, Villani E, Yoon KC, Jones L, Craig JP. TFOS DEWS II Diagnostic Methodology report. Ocul Surf. 2017 Jul;15(3):539-574. doi: 10.1016/j.jtos.2017.05.001. Epub 2017 Jul 20. PMID 28736342
- [Result] Aguilar AJ, Marquez MI, Albera PA, Tredicce JL, Berra A. Effects of Systane((R)) Balance on noninvasive tear film break-up time in patients with lipid-deficient dry eye. Clin Ophthalmol. 2014 Nov 25;8:2365-72. doi: 10.2147/OPTH.S70623. eCollection 2014. PMID 25473263
- [Result] Chiambaretta F, Doan S, Labetoulle M, Rocher N, Fekih LE, Messaoud R, Khairallah M, Baudouin C; HA-trehalose Study Group. A randomized, controlled study of the efficacy and safety of a new eyedrop formulation for moderate to severe dry eye syndrome. Eur J Ophthalmol. 2017 Jan 19;27(1):1-9. doi: 10.5301/ejo.5000836. Epub 2016 Jul 20. PMID 27445067
- [Result] Novack GD, Asbell P, Barabino S, Bergamini MVW, Ciolino JB, Foulks GN, Goldstein M, Lemp MA, Schrader S, Woods C, Stapleton F. TFOS DEWS II Clinical Trial Design Report. Ocul Surf. 2017 Jul;15(3):629-649. doi: 10.1016/j.jtos.2017.05.009. Epub 2017 Jul 20. PMID 28736344